CLINICAL TRIAL: NCT00145171
Title: Study of Orthostatic Changes Upon Apomorphine Dose Initiation in Late Stage Parkinson's Disease Patients. A Dose Escalation Study With a Double-Blind Placebo-Controlled Efficacy Determination at 4 Mg.
Brief Title: A Sub-Study With Patients in APO401 to Evaluate Adverse Events During Dose Introduction in Apomorphine-naïve Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APO303
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2002-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

INTERVENTIONS:
Drug: apomorphine HCl injection

SUMMARY:
APO303 is a sub-study of patients enrolled in APO401 (the long-term open label safety protocol) and was designed to evaluate adverse events, particularly blood pressure drops when standing up during first dose in patients who have not been exposed to apomorphine before.

DETAILED DESCRIPTION:
The primary objective of this study was to determine the electrocardiographic and orthostatic effects of apomorphine during controlled in-patient dose introduction in apomorphine-naïve late stage Parkinson's disease patients. Although safety observations represented the primary objective of the study, a control group was considered essential to properly interpret adverse events that occurred during dose titration. Additional data comparing the efficacy and safety of subcutaneous apomorphine, placebo and standard antiparkinson (anti-PD) therapy was derived from this experience.

This was a two-phase study that involved a controlled in-office dose titration phase followed by a 6-month outpatient open-label treatment phase. During the in-patient dose titration phase, subjects were evaluated on separate days for the response to single doses of medication administered during an observed "Off" event (defined as first "Off" event that occurs at least one hour after administration of the normal morning dose of oral antiparkinson medication). Evaluation of the acute response to oral anti-PD medication (Baseline) and to apomorphine dose escalation between 2 and 10 mg (Titration Visits) was conducted under unblinded conditions. At the 0.4-mL titration level, placebo was randomly introduced under double-blind crossover conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Adults of any age > 18.
2. Sex: Men and non-pregnant, non-lactating women.

   1. Women of childbearing potential must have had a negative serum (Beta HCG) pregnancy test within 14 days of the study start.
   2. Women of childbearing potential must have used an acceptable form of contraception
3. Patients with a clinical diagnosis of idiopathic Parkinson's disease, ie. not induced by drugs or caused by other diseases.
4. Patients classified as stage II - V of the Hoehn and Yahr scale for staging the severity of Parkinson's disease (Appendix 16.1.12.3).
5. Patients with refractory motor fluctuations of any frequency or duration. These included but are not necessarily limited to patients with the following symptoms:

   1. Immobility resulting from regular dose failures.
   2. Severe "Off" period discomfort.
   3. Nocturnal/early morning dystonias.
   4. Voiding dysfunctions.
   5. Swallowing difficulties associated with "Off" periods.
   6. "Off" period visual hallucinations.
   7. Severe biphasic dyskinesia.
6. Unless otherwise specified, enrolled patients must be on an optimally maximized oral therapy regimen. Optimized oral anti-PD medication included: levodopa/carbidopa in either immediate or delayed release forms, plus at least one other antiparkinson medication, which could include a direct acting oral dopamine agonist, a monoamine oxidase inhibitor (MAOB), or a catechol-O-methyltransferase inhibitor (COMT) for at least 30 days prior to enrollment into study.
7. Patients enrolled in APO401 who have completed initial baseline observations, but have not received apomorphine therapy as part of the APO401 protocol or at any other point in time.

Exclusion Criteria:

1. Patients with prior exposure to apomorphine, including prior participation in a Mylan sponsored study of subcutaneous apomorphine. Patients were enrolled in APO401 concurrently with APO303.
2. Patients who did not conform to all of the above inclusion criteria.
3. Patients under medical therapy for clinically significant psychoses or dementia.
4. Patients with a history of drug or alcohol dependency within one year prior to study enrollment.
5. Patients with unstable and clinically significant disease of cardiovascular (including orthostatic hypotension), hematologic (including Coombs' positive hemolytic anemia), hepatic, renal, metabolic, respiratory, gastrointestinal or endocrinological systems or neoplasm within the three months before the start of the study.
6. Patients on methyldopa therapy.
7. Patients with a history of true allergy to morphine or its derivatives, sulfur, sulfur containing medication, sulfites, trimethobenzamide or other anticholinergics.
8. Patients treated with other experimental agents within 30 days before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2001-02; Study Completion 2002-08

PRIMARY OUTCOMES:
Entire Study:
Adverse event assessments
For Crossover portion of placebo-controlled 4mg dose comparison:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) at 20 minutes after dosing

SECONDARY OUTCOMES:
1. Change in UPDRS Motor Score from pre-dose to 40 and 90 minutes after dosing;
2. Area under the curve (AUC) for UPDRS Motor Scores at 0, 20, 40 and 90 minutes;
3. Change in Dyskinesia Assessment at 0, 20, 40, and 90 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Will Sullivan, Study Director — Mylan Bertek Pharmaceuticals